CLINICAL TRIAL: NCT01665547
Title: Adding L-carnitine in Clomiphene Resistant Pco Improves the Quality of Ovulation and the Pregnancy Outcome,a Randomized Clinical Trial
Brief Title: Adding L-carnitine in Clomiphene Resistant Polycystic Ovary Improves the Quality of Ovulation and the Pregnancy Outcome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, alaa eldeen mahmoud ismail, assistant professor, Woman's Health University Hospital, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: lcpco
Record Dates: First submitted 2012-07-13; First posted 2012-08-15 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Treatment Resistant Disorders
Keywords: clomiphene resistant; pcos; induction of ovulation; l-carnitine
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- l-carnitine (Active Comparator): adding 3gm l-carnitine from day 1 to day 12 of induced the menstrual cycle by 50 mg clomiphene
  Interventions: Drug: l-carnitine

INTERVENTIONS:
Drug: l-carnitine — 3gm l-carnitine from day 1 to day 12 of the menstrual cycle
  Other Names: carivita,l-carnitol

SUMMARY:
Adding L-carnitine is more successful than clomiphene as a first line therapy for ovulation induction in women with clomiphene resistant PCOS

DETAILED DESCRIPTION:
Patients younger than 35 years, presenting with primary or secondary infertility following regular intercourse for at least 1 year and diagnosed with PCO according to Rotterdam's criteria who had received five unsuccessful clomiphene citrate-timed intercourse stimulation cycles were included.

ELIGIBILITY:
Inclusion Criteria:

* Patients younger than 35 years, presenting with primary or secondary infertility following regular intercourse for at least 1 year and diagnosed with PCO according to Rotterdam's criteria who had received five unsuccessful clomiphene citrate-timed intercourse stimulation cycles were included. The diagnosis was based on a complete history taking, physical examination and a paper documented complete infertility work-up within the previous 6 months, either conducted within the setting of the hospital or at a licensed infertility management clinic.

Exclusion Criteria:

* age more than 40 years,
* tubal,uterine or male factor infertility

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 157 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
ovulation induction | 0ne year
  is to study the efficacy of l-carnitine in inducing ovulation in clomiphene resistant pco

SECONDARY OUTCOMES:
pregnancy | 0ne year
  the occurrence of pregnancy and the rate of continuation of pregnancy till end of the first trimester

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Ismail, M.D, Principal Investigator — Women's Health Hospital